CLINICAL TRIAL: NCT04125953
Title: The Influence of Stochastic Modulated Vibrations on the Autonomic Nervous System of Breast Cancer Patients During Radiotherapy: a Randomized Clinical Trial
Brief Title: Stochastic Modulated Vibrations on Autonomic Nervous System of Breast Cancer Patients During Radiotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Nele, principal investigator, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2018/455
Record Dates: First submitted 2019-06-24; First posted 2019-10-14 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Autonomic Nervous System Imbalance; Psychological Distress; Cancer-related Pain; Breast Cancer Lymphedema; Quality of Life
MeSH Terms: conditions — Cancer Pain; Breast Cancer Lymphedema

STUDY DESIGN:
Intervention Model Description: randomized clinical trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): A 3 week intervention with Andullation will be performed, 3 times a week for 20 minutes after completion of the radiotherapy session
  Interventions: Device: Andullation
- Control (Placebo Comparator): This group will follow the same intervention protocol, but without the application of the Andullation technology
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Andullation — Andullation is a horizontal vibration technique with stochastically modulated vibrations, build-in in a mattress.
  Arms: Intervention
Other: Placebo — Placebo Andullation
  Arms: Control

SUMMARY:
The aim of this research is to study the influence of stochastic modulated vibrations on the autonomic nervous system of breast cancer patients during radiation therapy

DETAILED DESCRIPTION:
Since it is well known that breast cancer patients experience an important load of stress from diagnosis through treatment and throughout cancer survivorship (fear of cancer recurrence), this study focusses on activation the parasympathetic nervous system and making patients as comfortable as possible during treatment. The scope of this study is based on previous research, that has shown that controlling physical and psychological complications during treatment may have a positive (preventive) effect on late term and long-term quality of life and survival outcomes. Breast cancer patients will receive andullation during their irradiation period. The primary outcome measure of the autonomic nervous system is vagal nerve activity, a modulator of the parasympathetic nervous system. Secondary outcome measures are stress, pain and lymphedema.

ELIGIBILITY:
Inclusion Criteria:

* Histological proven breast cancer, following breast cancer surgery
* Starting with adjuvant radiation therapy for 3 weeks
* Minimum 18 years
* Medical record available and complete
* Supine lying on mattress for 20 minutes is possible
* Dutch, French or English

Exclusion Criteria:

* Severe neurological, orthopaedic or rheumatic disorders
* Cardiac disorders
* Early or synchronous malignancy
* Pregnancy or lactation
* Persons suffering from depression or illnesses which influence the mental health or wellbeing

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 130 (Estimated)
Dates: Start 2019-07-04 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
change in Heart Rate Variability (HRV) | through study completion, an average of 6 weeks
  a marker of the activity of your autonomic nervous system.

SECONDARY OUTCOMES:
change in Distress Thermometer | through study completion, an average of 6 weeks
  A questionnaire to evaluate in what extent you experience complaints like distress and anxiety, on a visual thermometer. By encircling the number most applicable for your situation, we can estimate how you are feeling at the moment. The scale ranges from 0-10 where 0 indicates a better and 10 indicates a worse outcome.
change in Brief Pain Inventory | through study completion, an average of 6 weeks
  This questionnaire was designed to investigate the extent of pain you experience as well as to examine the influence of it on your quality of life. The BPI includes four ratings of pain intensity (items 3-7), and seven other ratings on the impact of pain. Intensity is recorded on numerical scales from zero (no pain) to ten (pain as bad as you can imagine). Also, intensity is rated at the time of completing the questionnaires (pain now) as well as its worst, least, and average over the past day or week.
change in Numeric Pain Rating Scale | through study completion, an average of 6 weeks
  An 11-point scale for patient self-reporting of pain. The scale ranges from 0-10 where 0 indicates a better and 10 indicates a worse outcome.
change in Perometer results | through study completion, an average of 6 weeks
  A device measuring your arm circumferences with the use of infrared light. It is an efficient, safe, painless and reliable method to examine your arm circumferences.
change in Bioimpedance spectroscopy | through study completion, an average of 6 weeks
  By using bioimpedance, we will estimate your body fat, water and muscle content. You will stand on scale and hold on to a handgrip that is connected with the scale. A small current will determine your body composition. This is a painless and innocuous examination.
change in European Organization for Research and Treatment of Cancer 30-item core quality of life questionnaire (EORTC QLQ C-30) | through study completion, an average of 6 weeks
  A questionnaire designed to investigate the quality of life in cancer patients. The questionnaire assesses some domains of your quality of life that can possibly be influenced by your disease. The questionnaire consists of 3 different scales: Global Health Status (GHS), Functional Scale (FS) and Symptom Scale (SS). The answers of the FS and SS are scored on a Likert scale where lower scores indicate better outcomes.The GHS differs from the other scales by scoring on a 7-point Likert scale where lower scores display worse outcomes.
change in European Organization for Research and Treatment of Cancer 23-item quality of life questionnaire (EORTC QLQ BR23) | through study completion, an average of 6 weeks
  A questionnaire designed to investigate the quality of life in breast cancer patients. The questionnaire assesses some domains of your quality of life that can possibly be influenced by your disease. It consists of 23 questions to determine body image, sexual functioning, sexual enjoyment, future perspective, systemic therapy side effects, breast symptoms, arm symptoms and upset by hair loss assessed on a 4 point Likert scale where lower scores indicate better outcomes.
change in Pittsburgh Sleep Quality Index | through study completion, an average of 6 weeks
  A questionnaire that assesses your sleep quality, your sleep quantity and your sleep disturbance. The scale ranges from 0-21 where lower scores indicate better outcomes
change in Insomnia Severity Index | through study completion, an average of 6 weeks
  A questionnaire that assesses the severity, the nature and the impact of your insomnia over the past 2 - 4 weeks. The scale ranges from 0-28 where lower scores indicate better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Nele Adriaenssens, Prof. Dr., Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/53/NCT04125953/Prot_SAP_000.pdf